CLINICAL TRIAL: NCT03928600
Title: Labor Induction With a Combined Method (Pharmacologic and Mechanical): Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar De São João, E.P.E. (Other)
Responsible Party: Principal Investigator, Rita Polónia Valente, Principal Investigator, Centro Hospitalar De São João, E.P.E.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CES 171-17
Record Dates: First submitted 2019-03-04; First posted 2019-04-26 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Labor, Induced; Cervical Ripening
Keywords: induction of labor; cervical ripening; combined methods
MeSH Terms: interventions — Misoprostol; Dinoprostone; Mutagenesis, Insertional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combined method induction group (Experimental): * 25 micrograms misoprostol vaginal applied placed along with cervical Foley (team will repeat misoprostol application each 4 hours till 6 doses of misoprostol)
  * After 4 hours of last misoprostol initiate oxytocin.
  * Cervical Foley will be removed after 12h of placement or when fails out.
  Interventions: Combination Product: Cervical Foley combined with Misoprostol
- Current department guidelines group (Placebo Comparator): * Following current department guidelines, as usual, with the method considered more suitable.
  * If they opted for vaginal misoprostol, team will insert 25micrograms, repeat application 4/4h, until 150micrograms, after last misoprostol, wait 4 hours before initiating oxytocin.
  * If option is vaginal dinoprostone the insert of 10mg is removed after 24h in place.
  Interventions: Drug: Dinoprostone 10mg insert OR; Drug: Misoprostol

INTERVENTIONS:
Combination Product: Cervical Foley combined with Misoprostol — Placement of cervical Foley catheter along with application of vaginal misoprostol 25ug that will be repeated 4/4h until 150ug
  Arms: Combined method induction group
Drug: Dinoprostone 10mg insert OR — Application for 24h of Dinoprostone 10mg insert
  Arms: Current department guidelines group
Drug: Misoprostol — Application of vaginal misoprostol 25ug 4/4h until 150ug
  Arms: Current department guidelines group

SUMMARY:
Labor induction is a common pregnancy procedure worldwide. Both mechanical and pharmacologic agents are used for induction of labor. These agents reduce the incidence of cesarean delivery in women undergoing induction.

Opposite to old studies of cervical ripening, some recent studies have shown promise in reducing labor time and risk of cesarean delivery with combination methods. The effectiveness of this procedure is of major clinical importance and has a large impact in our quotidian practice.

The objective is to compare the effectiveness of a combined new method to current guidelines of our department

DETAILED DESCRIPTION:
We designed a randomized trial that will compare two groups: misoprostol-cervical Foley simultaneously and the current department guidelines (misoprostol alone/dinoprostone alone).

Inclusion criteria: full-term (≥ 37 weeks of gestation), singleton, vertex-

ELIGIBILITY:
Inclusion Criteria:

* full-term (≥ 37 weeks of gestation)
* singleton
* vertex-presenting gestations
* with no contraindication to vaginal delivery
* intact membranes
* Bishop score < 7 and cervical dilation ≤2 cm

Exclusion Criteria:

* contraindication for misoprostol
* history of previous caesarean
* rupture of membranes,
* fetal or maternal morbidities (fetal major abnormalities, FIGO definition of pathological CTG, HELLP syndrome, preeclampsia or hypertension with severe features, fetal growth restriction)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Time to delivery | 3 days
  Time to delivery

SECONDARY OUTCOMES:
cesarean delivery rate | 3 days
  cesarean delivery rate
time to active labor | 3 days
  defined as dilation of 6 cm or greater
rate of delivery within 12 hours | 12 hours
  rate of delivery within 12 hours
rate of delivery within 24 hours | 24 hours
  rate of delivery within 24 hours
mean of maternal length of stay | average 3 days
  induction to discharge
indication for cesarean delivery | 3 days
  indication for cesarean delivery
composite maternal morbidity outcome | 6 weeks
  third- or fourth-degree perineal laceration, blood transfusion, chorioamnionitis, endometritis, wound infection, venous thromboembolism, hysterectomy, intensive care unit admission or death.
composite of neonatal morbidities | 30 days
  SDR, neonatal sepsis, blood transfusion, encephalopathy hypoxic-ischemic, intraventricular hemorrhage of grade III/IV

CONTACTS AND LOCATIONS:
Overall Officials: Rita P Valente, MD, Principal Investigator — Centro Hospitalar São João, Porto
Locations (1):
- Centro Hospitalar São João, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Informed Consent Form, Statistical Analysis Plan
Supporting Information: Study Protocol, SAP, ICF
Time Frame: no ending
Access Criteria: Researchers who provide a methodologically sound proposal.